CLINICAL TRIAL: NCT05332392
Title: Clinical Performance of Masimo INVSENSOR00040
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CIP-1019
Record Dates: First submitted 2022-04-11; First posted 2022-04-18 (Actual); Results first posted 2024-02-28 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-01

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- INVSENSOR00040 (Experimental): All subjects who are enrolled into the test group and participate in data collection receive the noninvasive INVSENSOR00040 device.
  Interventions: Device: INVSENSOR00040

INTERVENTIONS:
Device: INVSENSOR00040 — Noninvasive wearable health monitoring device

SUMMARY:
This study is designed to compare the accuracy of a noninvasive measurement of oxygen saturation and pulse rate to reference values obtained by a laboratory blood gas analyzer and a standard of care EKG monitor.

Study procedures follow ISO-80601-2-61:2011 standard requirements for basic safety and essential performance of pulse oximeter equipment. Arterial blood samples will be collected from subjects while undergoing a controlled desaturation procedure wherein the concentration of oxygen inhaled is slowly reduced until the subject's arterial oxygen concentration is approximately 70%.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 to 50 years of age.
* Subject weighs a minimum of 110 lbs.
* Subject has a hemoglobin value ≥ 11 g/dL.
* Subject's baseline heart rate is ≥ 45 bpm and ≤ 85 bpm.
* Subject's CO value is ≤ 3.0% FCOHb.
* Subject's blood pressure: Systolic BP ≤ 140 mmHg and ≥ 90 mmHg, Diastolic BP ≤ 90 mmHg and ≥ 50 mmHg, and if systolic BP is lower than 100 mmHg and/or diastolic BP is lower than 60 mmHg, subject passes an orthostatic blood pressure test.
* Subject is able to read and communicate in English and understands the study and the risks involved.

Exclusion Criteria:

* Subject whose skin is not intact and/or has tattoos in the area of device placement (e.g., wrist).*
* Subject is pregnant.
* Subject has a BMI > 35.
* Subject has a history of fainting (vasovagal syncope), blacking out or losing consciousness during or after a blood draw, or has a fear of blood draws.
* Subject has open wounds, inflamed tattoos or piercings, and/or has any visible healing wounds that a medical professional determines may place them at an increased risk for participation.*
* Subject has known drug or alcohol abuse.
* Subject uses recreational drugs.*
* Subject experiences frequent or severe headaches and/or migraine headaches, migraine auras, altitude sickness, and/or headaches accompanied by visual changes or sensitivity to light or sound.
* Subject has experienced a concussion or head injury with loss of consciousness within the past 12 months.
* Subject has any history of a stroke, myocardial infarction (heart attack), and/or seizures.
* Subject has any chronic bleeding disorder (e.g. hemophilia).
* Subject has taken anticoagulant medication within the past 30 days (excluding nonsteroidal anti-inflammatory drugs (NSAIDS)).
* Subject has donated blood within the past 4 weeks.
* Subject has Wolff-Parkinson-White Syndrome or Stokes-Adams Syndrome.
* Subject has any symptomatic cardiac dysrhythmia (e.g. atrial fibrillation) and has not received clearance from their physician to participate.
* Subject has a known neurological and/or psychiatric disorder (e.g. schizophrenia, bipolar disorder, multiple sclerosis, Huntington's disease) that interferes with the subject's level of consciousness.*
* Subject has taken opioid pain medication 24 hours before the study.
* Subject has any active signs and/or symptoms of infectious disease (e.g. hepatitis, HIV, tuberculosis, flu, malaria, measles, etc.).*
* Subject is taking medications known to treat any type of infectious disease.
* Subject has either signs or history of peripheral ischemia or carpal tunnel syndrome.
* Subject has had invasive surgery within the past year, including but not limited to major dental surgery, appendectomy, plastic surgery, jaw surgery, major ENT surgery, major abdominal and/or pelvic surgery, heart surgery, or thoracic surgery.*
* Subject has symptoms of congestion, head cold, or other illnesses.
* Subject has been in a severe car accident(s) or a similar type of accident(s) requiring hospitalization within the past 12 months.
* Subject has any cancer or history of cancer (not including skin cancer).*
* Subject has chronic unresolved asthma, lung disease (including COPD) and/or respiratory disease.
* Subject is allergic to lidocaine, chlorhexidine, latex, adhesives, or plastic.
* Subject has a heart condition, insulin-dependent diabetes, or uncontrolled hypertension.
* Subject has delivered vaginally, has had a pregnancy terminated, a miscarriage with hospitalization, or had a C-section within the past 6 months.
* Subject intends on participating in any heavy lifting, repetitive movement of their wrist (including riding a motorcycle, tennis), exercise (working out, riding a bike, riding a skateboard, etc.), or any activity that will put additional stress on the wrist within 24 hours following a study that involves an arterial line.
* Subject has any medical condition which in the judgment of the investigator and/or medical staff, renders them ineligible for participation in this study or subject is deemed ineligible by the discretion of the investigator/study staff.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2022-04-14 (Actual); Primary Completion 2023-04-13 (Actual); Study Completion 2023-04-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Masimo Corporation, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | INVSENSOR00040
Started | 90
Completed | 46
Not Completed | 44
Not completed — Did not meet inclusion criteria | 25
Not completed — Principal Investigator's decision | 17
Not completed — Adverse Event | 1
Not completed — Subject's decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | INVSENSOR00040
Number analyzed (Participants) | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 46
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: African American | 15
  Ethnicity: Asian or Pacific Islander | 9
  Ethnicity: African American & Asian or Pacific Islander | 1
  Ethnicity: Hispanic | 9
  Ethnicity: White | 11
  Ethnicity: White & Native American | 1
Region of Enrollment [Number; unit: participants]
  United States | 46

OUTCOME MEASURES:

1. Primary Outcome: Oxygen Saturation (SpO2) Accuracy of INVSENSOR00040
Description: SpO2 performance will be determined by calculating the arithmetic root square mean (ARMS) value through the comparison of the noninvasive SpO2 measurement obtained from INVSENSOR00040 to the arterial oxygen saturation (SaO2) value obtained from a reference blood sample.
  The square root of the sum of the squares of bias and precision is computed as the ARMS Error Value.
  The desaturation range over which the accuracy is performed is 70-100%.
Time Frame: 1-5 hours
Population: Data from 13 subjects was excluded due to desaturation procedural error. Data from 1 subject was excluded due to missing data and evidence of noise interference that did not allow for the comparison of the dataset.
  Data from 1 subject was excluded because the subject complained of discomfort at the early part of the desaturation procedure and therefore was unable to desaturate to below 90% SaO2.
Measure: Number; unit: % of oxygen saturated hemoglobin
Arm/Group | INVSENSOR00040
Number analyzed (Participants) | 31
% of oxygen saturated hemoglobin | 1.62

2. Primary Outcome: Pulse Rate (PR) Accuracy of INVSENSOR00040
Description: Pulse Rate (PR) performance will be determined by calculating the ARMS value through the comparison of the PR values obtained from INVSENSOR00040 to the heart rate (HR) values obtained from a reference standard of care EKG monitor.
  The square root of the sum of the squares of bias and precision is computed as the ARMS Error Value.
  The PR/HR range over which the accuracy is calculated is determined by convenience sampling in a generally healthy population undergoing a desaturation procedure.
Time Frame: 1-5 hours
Population: Data from 13 subjects excluded due to desaturation procedural error. Data from 1 subject excluded due to missing data & evidence of noise interference that did not allow for the comparison of the dataset.
  Data from 1 subject excluded because subject complained of discomfort at early part of desaturation procedure, therefore was unable to desaturate to below 90% SaO2.
  Data from 2 subjects excluded for no valid PR & ECG HR pair, because ECG HR data was not recorded in the server properly.
Measure: Number; unit: beats per minute
Arm/Group | INVSENSOR00040
Number analyzed (Participants) | 29
beats per minute | 1.29

ADVERSE EVENTS:
Time Frame: 1 to 5 hours
Arm/Group | INVSENSOR00040
All-Cause Mortality (participants affected / at risk) | 0/46
Serious Adverse Events (participants affected / at risk) | 0/46
Other Adverse Events (participants affected / at risk) | 4/46
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | INVSENSOR00040 (N=46)
Unilateral temporal headache (Injury, poisoning and procedural complications) | 1 (1)
Lightheadedness (Injury, poisoning and procedural complications) | 1 (1)
Swelling/Tenderness at arterial line site (Injury, poisoning and procedural complications) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-14): https://cdn.clinicaltrials.gov/large-docs/92/NCT05332392/Prot_SAP_000.pdf